CLINICAL TRIAL: NCT00741026
Title: A Double-blind, Placebo-controlled, Crossover Study Examining the Acute Effects of Olanzapine on Plasma Leptin, Glucose Tolerance and Free Fatty Acids in Healthy Volunteers
Brief Title: A Crossover Study of the Acute Effects of Olanzapine in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: American Medical Association (Other)
Responsible Party: Principal Investigator, Vance L. Albaugh, MD/PhD Student, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 28230
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Insulin Resistance; Diabetes Mellitus
Keywords: Insulin Resistance; Diabetes mellitus; Antipsychotic
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus | interventions — Olanzapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Olanzapine (Experimental): Olanzapine 10mg po daily x 3 days
  Interventions: Drug: Olanzapine 10 mg po qhs for 3 days

INTERVENTIONS:
Drug: Olanzapine 10 mg po qhs for 3 days — (1) 10 mg tablets administered orally before bed for three consecutive evenings (Total Dose = 30 mg, 3 tablets)
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Placebo — (1) placebo tablets administered orally before bed for three consecutive evenings (Total Dose = 3 tablets)
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this clinical research study is to examine the acute hormonal and metabolic effects of the drug olanzapine, as well as appetite effects, in healthy volunteers. The hypotheses to be tested are that: (1) Olanzapine rapidly attenuates plasma leptin and (2) rapidly alters glucose tolerance in healthy volunteers. These questions will be answered by having volunteers undergo two glucose tolerance tests in a crossover study design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer
* Body Mass Index of 18.5-25 kilograms per square meter
* Must be able to swallow tablets
* Able to give informed consent

Exclusion Criteria:

* Any DSM-IV TR Axis I psychiatric disorder (except nicotine dependence)
* Presence of any medical disorder that may confound the assessment of relevant biologic measures, including: significant organ system dysfunction, metabolic diseases, type 1 diabetes mellitus, type 2 diabetes mellitus, pregnancy, endocrine disease, coagulopathy, clinically significant anemia, or acute infection
* Subjects who have taken any antipsychotic medication within the last 6 months
* Personal or family history of seizures and/or cardiac arrhythmias

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Singareddy, M.D., Study Director — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center; Vance L Albaugh, M.D., Ph.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Albaugh VL, Henry CR, Bello NT, Hajnal A, Lynch SL, Halle B, Lynch CJ. Hormonal and metabolic effects of olanzapine and clozapine related to body weight in rodents. Obesity (Silver Spring). 2006 Jan;14(1):36-51. doi: 10.1038/oby.2006.6. PMID 16493121
- [Background] Albaugh VL, Judson JG, She P, Lang CH, Maresca KP, Joyal JL, Lynch CJ. Olanzapine promotes fat accumulation in male rats by decreasing physical activity, repartitioning energy and increasing adipose tissue lipogenesis while impairing lipolysis. Mol Psychiatry. 2011 May;16(5):569-81. doi: 10.1038/mp.2010.33. Epub 2010 Mar 23. PMID 20308992
- [Background] Albaugh VL, Vary TC, Ilkayeva O, Wenner BR, Maresca KP, Joyal JL, Breazeale S, Elich TD, Lang CH, Lynch CJ. Atypical antipsychotics rapidly and inappropriately switch peripheral fuel utilization to lipids, impairing metabolic flexibility in rodents. Schizophr Bull. 2012 Jan;38(1):153-66. doi: 10.1093/schbul/sbq053. Epub 2010 May 21. PMID 20494946
- [Result] Albaugh VL, Singareddy R, Mauger D, Lynch CJ. A double blind, placebo-controlled, randomized crossover study of the acute metabolic effects of olanzapine in healthy volunteers. PLoS One. 2011;6(8):e22662. doi: 10.1371/journal.pone.0022662. Epub 2011 Aug 9. PMID 21857944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 individuals were screened between July 2008 and June 2009, and of those individuals 15 subjects were eligible based on inclusion/exclusion criteria.
Pre-assignment Details: Only individuals that met inclusion/exclusion criteria were allowed to participate in the study. Of the 42 individuals screened, only 15 met criteria and were interested in taking part in the study. There was a minimum 2 week washout period in between treatment arms (i.e. placebo vs active compound).
Groups:
- Placebo / Olanzapine: Participants that were randomized to Placebo (Sugar Pill) treatment for three days and then a washout period of at least two weeks but not more than 4 weeks before Olanzapine treatment, 10 mg olanzapine by mouth at bedtime for three consecutive nights.
  OR
  Participants that were randomized to Olanzapine, 10 mg olanzapine by mouth at bedtime for three consecutive nights before a washout period of at least two weeks but not more than 4 weeks before Placebo treatment (Sugar Pill) for three days.
  Randomization information not available.
Period: Overall Study
Arm/Group | Placebo / Olanzapine
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo / Olanzapine: Participants that were randomized to Placebo (Sugar Pill) treatment for three days and then a washout period of at least two weeks but not more than 4 weeks before Olanzapine treatment, 10 mg olanzapine by mouth at bedtime for three consecutive nights.
  OR
  Participants that were randomized to Olanzapine, 10 mg olanzapine by mouth at bedtime for three consecutive nights before a washout period of at least two weeks but not more than 4 weeks before Placebo treatment (Sugar Pill) for three days.
Arm/Group | Placebo / Olanzapine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Plasma Leptin
Description: Leptin following placebo or olanzapine treatment
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
ng/ml | 6.8 (1.3) | 8.4 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Olanzapine; Test type: Superiority or Other; p = 0.0203, Wilcoxon Signed-rank

2. Primary Outcome: Oral Glucose Tolerance
Description: Oral Glucose Tolerance
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: min*mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
min*mg/dl | 2808 (474) | 3984 (444)
Statistical Analysis 1: Comparison: Placebo vs Olanzapine; Test type: Superiority or Other; p = 0.0105, Wilcoxon Sign-rank

3. Primary Outcome: Plasma Free Fatty Acid
Description: Plasma Free Fatty Acid
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mM | 0.38 (0.06) | 0.26 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Olanzapine; Test type: Superiority or Other; p = 0.0166, Wilcoxon Sign-rank

4. Secondary Outcome: HDL Cholesterol
Description: HDL Cholesterol
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mg/dl | 54.2 (4.7) | 48.9 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Olanzapine; Test type: Superiority or Other; p = 0.0184, Wilcoxon Sign-rank

5. Secondary Outcome: Triglycerides
Description: Triglycerides
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mg/dl | 88.9 (10.1) | 108.2 (11.6)
Statistical Analysis 1: Comparison: Placebo vs Olanzapine; Test type: Superiority or Other; p = 0.0170, Wilcoxon Sign-rank

6. Secondary Outcome: LDL Cholesterol
Description: LDL Cholesterol
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mg/dl | 82.7 (6.6) | 81.7 (7.8)

7. Secondary Outcome: Total Cholesterol
Description: Total Cholesterol
Time Frame: 3 Days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mg/dl | 156.8 (9.1) | 152.6 (10.1)

8. Secondary Outcome: Body Weight
Description: Body Weight
Time Frame: 3 Days
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
kg | 68.2 (2.9) | 68.9 (3.0)

9. Secondary Outcome: BMI
Description: BMI
Time Frame: 3 Days
Measure: Mean (Standard Error); unit: kg / m2
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
kg / m2 | 23.0 (0.5) | 23.0 (0.6)

10. Secondary Outcome: Heart Rate
Description: Heart Rate
Time Frame: 3 Days
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
beats per minute | 69.9 (2.6) | 67.6 (3.5)

11. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood Pressure
Time Frame: 3 Days
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mmHg | 113.3 (2.8) | 111.7 (3.1)

12. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood Pressure
Time Frame: 3 Days
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Olanzapine
Number analyzed (Participants) | 15 | 15
mmHg | 68.3 (2.0) | 69.5 (1.8)

ADVERSE EVENTS:
Groups:
- Placebo: Placebo : (1) placebo tablets administered orally before bed for three consecutive evenings (Total Dose = 3 tablets)
Arm/Group | Placebo | Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
One episode of orthostatic hypotension requiring unblinding. One individual with emesis after glucose challenge and that individual's glucose tolerance data were unavailable analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No